CLINICAL TRIAL: NCT06897995
Title: The Effects of Aerobic Exercise on Aerobic Fitness and Platelet Mitochondrial Bioenergetics
Brief Title: Aerobic Exercise on Platelet Mitochondrial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jong-Shyan Wang, Prof, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202300538B0
Record Dates: First submitted 2025-03-19; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-02

CONDITIONS: Sedentary Lifestyle; Aerobic Exercise
Keywords: mitochondrial respiration; oxidative stress; physical exercise; thrombocytes
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exercise; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Circuit training group (Experimental)
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION
- Cycle ergometer group (Active Comparator)
  Interventions: Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION

INTERVENTIONS:
Other: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — Participants in the exercise groups were trained five times a week for six weeks. The regimen began with a 5-min warm-up and ended with a 5-min cool-down, both at 40% of heart rate reserved (HRR). The circuit training participants were trained for three bouts of 10-min moderate-intensity exercise (60% of HRR) with 1-min rest intervals at a stationary ergometer, a rowing machine, and an elliptical trainer, respectively. The cycling training group was trained on an ergometer for three bouts of 10-min cycling on a stationary ergometer.

SUMMARY:
This study explores how exercise affects blood platelets and their role in clotting. Regular exercise can influence how efficiently clots form in the body. Intense exercise tends to increase platelet activity and the expression of certain molecules on their surface, while moderate exercise can decrease this activity. Since platelets are responsible for blood clotting, understanding how they function can be crucial.

Understanding Platelets:

Platelets are blood cells that help in clotting. The mitochondria within platelets help regulate their function. If these mitochondria don't work properly, it can lead to issues with clotting. By examining how exercise changes platelet mitochondria, the investigators can potentially identify important markers for health and disease progression.

Study Design:

This study compares two types of exercise routines: circuit training and stationary bicycle training.

Participants will be randomly assigned to one of the two groups:

Circuit Training Group: This involves moving through different exercise stations within a set time, targeting various body parts. It's tailored for those who might find regular exercise challenging, helping to reduce fatigue in any single area and improve overall fitness.

Bicycle Training Group: This involves exercising on a stationary bike. Both exercise groups will engage in high-intensity interval training for about 40 minutes, five times a week, over six weeks.

Assessment: Participants will undergo tests to measure endurance and physical function.

Blood Sampling: Blood will be drawn before and after the exercise tests, with 20 milliliters taken from the arm vein. Blood samples will also be collected at the start and end of a 6-week intervention, totaling 80 milliliters throughout the study. This helps the investigators analyze how platelets are affected by exercise.

This study is designed to help the investigators better understand how different types of exercise can benefit platelet function and overall health. Participanting in this research could contribute to the knowledge about how could exercise influence blood clotting and related health conditions. Participants' involvement will include exercise routines or maintaining your current lifestyle, along with simple blood tests. Participation is highly valuable and can help pave the way for new health insights and treatments.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign a written informed consent form.
* Ages 18 to 28.
* No regular exercise habit (defined as exercising 2 times a week or less, for 60 minutes or less each time, for over a year).

Exclusion Criteria:

* Overweight (BMI > 24) or underweight (BMI < 19).
* Smoked within the past year, or consumed alcohol in the past month exceeding 60 grams of alcohol per occasion.
* Having metabolic, circulatory, respiratory, or immune-related diseases or risk factors such as diabetes, hyperlipidemia, hypertension, heart disease, clotting disorders, asthma, allergies, autoimmune diseases, etc.
* Long-term use of any nutritional supplements or medications (e.g., vitamins, pain relievers, aspirin, traditional Chinese medicine).
* Significant knee injuries within the past year (e.g., ligament damage, fractures).
* Students and laboratory staff taught, assessed, evaluated, tested, or appraised by the principal investigator of this study.

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Platelet mitochondrial respiration | baseline and 2 days upon the completion of the 6-week intervention
  The mitochondrial OXPHOS and ET capacities in platelets were analyzed.
Cardiopulmonary fitness | baseline and 2 days upon the completion of the 6-week intervention
  Graded Exercise Test was performed on an ergometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided